CLINICAL TRIAL: NCT01481727
Title: Exacerbation's Prevention in Patients With COPD in GOLD IV Stage (Very Severe) With Non Invasive Mechanical Ventilation
Brief Title: Exacerbation Prevention GOLD IV COPD With Non Invasive Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Alejandra Ramirez Venegas, Head of COPD Clinic, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: C-18-10NIRD
Record Dates: First submitted 2011-10-20; First posted 2011-11-29 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: acute exacerbation of COPD number; acute exacerbation of COPD severity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cpap sham (Placebo Comparator): non invasive mechanical ventilation type cpap sham manoeuver
  Interventions: Device: BiPAP Pro 2, Phillips Respironics; Device: CPAP sham
- high-intensity NIMV (Active Comparator): Non-invasive mechanical ventilation, biPAP modality, with high-intensity IPAP (>18cmH2O)
  Interventions: Device: BiPAP Pro 2, Phillips Respironics

INTERVENTIONS:
Device: BiPAP Pro 2, Phillips Respironics — mechanical ventilation type bilevel at high intensity (>18mmHg) for at least six hours, nocturnal ventilation.
  Other Names: high intensity non invasive ventilation; high intensity bilevel
Device: CPAP sham — CPAP sham maneuver (IPAP less or equal to 4cmH2O)
  Other Names: placebo CPAP; sham non invasive ventilation
  Arms: cpap sham

SUMMARY:
The purpose of this study is to evaluate the efficacy of high-intensity non invasive mechanical ventilation (during one year to reduce the severity and frequency of acute exacerbation of chronic obstructive pulmonary disease (AECOPD) in patients with frequent AECOPD (frequent exacerbations defined more two or more AECOPD) and in GOLD IV stage (very severe COPD). The design is a randomised, double blind and controled with placebo (sham maneuver) clinical trial.

DETAILED DESCRIPTION:
Background:

* There are many previous studies (no controlled trials or observational studies)that demonstrated minimal benefits (on gas exchange and marginal effect over exacerbations frequency) with the use of non invasive mechanical ventilation, in BiPAP modality with IPAP pressures <18H2ocm (low intensity), in COPD patients.
* In subsequent years there were controled trials that concluded that there was no benefits with the use of non invasive mechanical ventilation on BiPAP mode in COPD patients ( It should be mentioned that in most trials were used low inspiratory pressure levels, that is called low-intensity non invasive mechanical ventilation).
* However, there are other recent studies that described some benefits of high intensity Bilevel modality of non invasive mechanical ventilation (inspiratory pressures >18cmH2O) specially on gas exchange, quality of life and functional status.
* There are some issues that do not yet have a clear answer like the optimal inspiratory pressure (IPAP) or the ventilation modality (BIPAP or other) to obtain the maximal benefit on COPD patients. Additionally, is not clear also if the use of non invasive mechanical ventilation on COPD patients helps to reduce the frequency and severity of acute exacerbations of COPD (AECOPD).

This study have some characteristics that are different to the previous reports:

* The inclusion of patients with frequent exacerbations phenotype (and therefore worst prognosis patients)that there are no included in previous trials
* The intervention maneuver that is bilevel modality of non invasive mechanical ventilation at hig-intensity pressure (>18H2Ocm and <24H2Ocm)
* The use of placebo maneuver (CPAP "Sham")
* The home titration in three phases, over a week
* The long-term use of the intervention and sham maneuver

ELIGIBILITY:
Inclusion Criteria:

* Clinical and spirometric diagnosis for COPD (FEV1/FVC <70%)
* Clinical phenotype of frequent exacerbations
* Must sign the informed consent
* Former smokers
* Stable COPD
* FEV1 <35%
* Optimal medical treatment

Exclusion Criteria:

* OSAS diagnosis
* Other indications for non invasive mechanical ventilation
* Arterial pressure for dioxide carbon >45mmHg
* Lung cancer
* Impossibility for doing spirometry or going to the medical visits
* Be included in another study

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
acute exacerbations of Chronic Obstructive Pulmonary Disease frequency | 1 year
  It will be calculated the exacerbation/year-patien rate and will be compared between groups
acute exacerbation of chronic obstructive pulmonary disease severity | 1 year
  It will be measured the rate of AECOPD with hospitalary and Intensive Care Unity requirement

SECONDARY OUTCOMES:
lymphocyte subpopulations Th-1 and Th-17 | 1 year
  It will be measured the lymphocyte subpopulations like Th-1 and Th-17
six-minute walking test | 1 year
Forced expiratory volume in first second (FEV1) and forced expiratory capacity | 1 year
Maximal inspiratory pressure and maximal expiratory pressure | 1 año
gas exchange response (carbon and oxygen dioxide arterial pressure) | 1 year
Health related quality of life | one year
anxiety and depression measures (HAD and Beck Questionnaires) | one year
echocardiographic parameters | one year
survival | one year
IL-1 and IL-6 cytokines | one year
  it will be measured the level of interleukines 1 and 6(IL-1 and IL-6)

CONTACTS AND LOCATIONS:
Overall Officials: RAUL HUMBERTO SANSORES MARTINEZ, MMS and MD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- National Institute of Respiratory Diseases, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] McEvoy RD, Pierce RJ, Hillman D, Esterman A, Ellis EE, Catcheside PG, O'Donoghue FJ, Barnes DJ, Grunstein RR; Australian trial of non-invasive Ventilation in Chronic Airflow Limitation (AVCAL) Study Group. Nocturnal non-invasive nasal ventilation in stable hypercapnic COPD: a randomised controlled trial. Thorax. 2009 Jul;64(7):561-6. doi: 10.1136/thx.2008.108274. Epub 2009 Feb 12. PMID 19213769
- [Background] Clini E, Sturani C, Rossi A, Viaggi S, Corrado A, Donner CF, Ambrosino N; Rehabilitation and Chronic Care Study Group, Italian Association of Hospital Pulmonologists (AIPO). The Italian multicentre study on noninvasive ventilation in chronic obstructive pulmonary disease patients. Eur Respir J. 2002 Sep;20(3):529-38. doi: 10.1183/09031936.02.02162001. PMID 12358325
- [Background] Casanova C, Celli BR, Tost L, Soriano E, Abreu J, Velasco V, Santolaria F. Long-term controlled trial of nocturnal nasal positive pressure ventilation in patients with severe COPD. Chest. 2000 Dec;118(6):1582-90. doi: 10.1378/chest.118.6.1582. PMID 11115443
- [Background] Lin CC. Comparison between nocturnal nasal positive pressure ventilation combined with oxygen therapy and oxygen monotherapy in patients with severe COPD. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):353-8. doi: 10.1164/ajrccm.154.2.8756806.
- [Background] Windisch W, Haenel M, Storre JH, Dreher M. High-intensity non-invasive positive pressure ventilation for stable hypercapnic COPD. Int J Med Sci. 2009;6(2):72-6. doi: 10.7150/ijms.6.72. Epub 2009 Feb 27. PMID 19277252
- [Background] Dreher M, Storre JH, Schmoor C, Windisch W. High-intensity versus low-intensity non-invasive ventilation in patients with stable hypercapnic COPD: a randomised crossover trial. Thorax. 2010 Apr;65(4):303-8. doi: 10.1136/thx.2009.124263. PMID 20388753
- [Background] Windisch W, Kostic S, Dreher M, Virchow JC Jr, Sorichter S. Outcome of patients with stable COPD receiving controlled noninvasive positive pressure ventilation aimed at a maximal reduction of Pa(CO2). Chest. 2005 Aug;128(2):657-62. doi: 10.1378/chest.128.2.657. PMID 16100151
- [Background] Budweiser S, Hitzl AP, Jorres RA, Heinemann F, Arzt M, Schroll S, Pfeifer M. Impact of noninvasive home ventilation on long-term survival in chronic hypercapnic COPD: a prospective observational study. Int J Clin Pract. 2007 Sep;61(9):1516-22. doi: 10.1111/j.1742-1241.2007.01427.x. PMID 17686094